CLINICAL TRIAL: NCT00249678
Title: Behavioral Therapy Development for Methamphetamine Abuse
Brief Title: Behavioral Therapy Development for Methamphetamine Abusers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left the institution before enrolling any participants
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Purpose: Treatment
Other Study IDs: NIDA-18075-1; R21DA018075 (NIH); R21-18075-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: The Study Was Designed to Develop a Cognitive Behavioral Approach to Treating Methamphetamine Abuse in HIV Primary Care Settings
Keywords: Behavior Therapy; methamphetamine
MeSH Terms: interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is...to assess whether placing a substance abuse intervention for HIV+ methamphetamine users within an HIV medical care setting improves rates of follow-up on referral to treatment by primary care physicians; reduces drug use and sexual risk behaviors more than treatment-as-usual; and increases rates of adherence to HIV medication regimens.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-seropositive, GBM receiving medical treatment for HIV for at least 30 days prior to signing informed consent at the UCLA CARE clinic, aged 18-65
2. Willing to give informed consent and comply with study procedures;
3. Willing to provide consent to contact treating physicians and pharmacies to assess adherence to HIV medications;
4. Diagnosed with current methamphetamine abuse as determined by MINI; and
5. Interested in seeking treatment for their methamphetamine abuse and in participating in this research project.

Exclusion Criteria:

1. Unwilling to give, or withdrawal of, informed consent;
2. Inability to understand nature of study;
3. A psychiatric condition that, in the principal investigator's judgment, warrants additional intervention to ensure participant safety (e.g., meets DSM-IV-TR criteria for current bipolar disorder or a psychotic disorder);
4. Current suicidal ideation or suicide attempt within the past 3 months; and
5. Concurrent dependence on opiates, alcohol, or benzodiazepines as determined by MINI.
6. Total lack of any type of healthcare coverage. These potential participants will be given low-fee treatment referrals.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-09 (Estimated); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Craving
Medication compliance
Addiction severity
Psychiatric interview
Sex-risk behavior

SECONDARY OUTCOMES:
Depression
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: James Peck, Other, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - UCLA, Integrated Substance Abuse Programs, Los Angeles, California
  - UCLA CARE Clinic, Los Angeles, California